CLINICAL TRIAL: NCT06755541
Title: An Open Label Long-Term Study to Evaluate the Safety and Tolerability of Fenofibrate in Combination With Ursodeoxycholic Acid in Subjects With Primary Biliary Cholangitis (PBC)
Brief Title: Fenofibrate in Combination With Ursodeoxycholic Acid in Primary Biliary Cholangitis: a Real World Study
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Xijing Hospital of Digestive Diseases (Other)
Responsible Party: Principal Investigator, Han Ying, Professor, Xijing Hospital of Digestive Diseases
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY20222274-C-1-1
Record Dates: First submitted 2024-12-24; First posted 2025-01-01 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Primary Biliary Cholangitis (PBC)
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — Fenofibrate; Ursodeoxycholic Acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- fenofibrate (Experimental): Experimental: Fenofibrate 200 mg Capsules
  Interventions: Drug: Fenofibrate in Combination With Ursodeoxycholic Acid

INTERVENTIONS:
Drug: Fenofibrate in Combination With Ursodeoxycholic Acid — Experimental: Fenofibrate 200 mg Capsules

SUMMARY:
An Open Label Long-Term Study to Evaluate the Safety and Tolerability of Fenofibrate in Combination with Ursodeoxycholic Acid in Subjects with Primary Biliary Cholangitis (PBC)

ELIGIBILITY:
Inclusion Criteria:

1. Must have given written informed consent (signed and dated)
2. Completed in a PBC study with fenofibrate(NCT05751967)
3. Females of reproductive potential must use at least one barrier contraceptive and a second effective birth control method during the study and for at least 90 days after the last dose. Male subjects who are sexually active with female partners of reproductive potential must use barrier contraception and their female partners must use a second effective birth control method during the study and for at least 90 days after the last dose

Exclusion Criteria:

1. Treatment-related adverse event (AE) leading to study drug discontinuation in a previous PBC study with seladelpar
2. A medical condition, other than PBC, that in the Investigator's opinion would preclude full participation in the study or confound its results

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-01-30 (Actual); Primary Completion 2035-12 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Treatment emergent adverse events (TEAEs) | Through study completion, up to 120 Months

SECONDARY OUTCOMES:
Death | 120 months
  Occurrence of overall death
Liver transplantation | 120 months
  Occurrence of overall liver transplantation
Normalization of ALP | 120 months
  Proportion of subjects with normalization of ALP

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing hospital, Xi'an, Shaanxi, China